CLINICAL TRIAL: NCT03890601
Title: Domain 1 of β2-Glycoprotein 1 Autoantibodies and Thrombin Generation Capacity in Patients With Antiphospholipid Antibodies
Brief Title: New Biological Tests in Patients With Antiphospholipid Antibodies
Acronym: LYON SAPL
Status: Recruiting | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL18_0522; 2018-A03020-55 (Other: ID-RCB)
Record Dates: First submitted 2019-02-28; First posted 2019-03-26 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Antiphospholipid Syndrome
MeSH Terms: conditions — Antiphospholipid Syndrome | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — A single 15 mL blood draw is planned for this study, as follow: 10 mL citrated tube (2 tubes) for activated Partial Prothrombin Time (APTT), Prothrombin Time (PT), D-Dimers, Lupus anticoagulant (LA), Anti-cardiolipin antibodies (aCL), Anti-β2 Glycoprotein1 antibodies (aβ2GP1), Antibodies to Domain 1 (Dm1) of β2-Glycoprotein 1 (aβ2GP1-dm1) and Thrombin Generation Assay (TGA ) ; and 5 mL ethylenediaminetetraacetic acid (EDTA) tube for blood count. During a follow up visit, a 5 ml citrated tube and a 5 mL EDTA tube are collected from each patient for their routine laboratory evaluation. One additional citrated tube will be required to measure thrombin generation and aβ2GP1-dm1. Platelet-poor plasmas will be prepared by double centrifugation at 2 500 g for 15 minutes at room temperature and then all citrated plasma samples will be stored at -80°C. At the end of the study, the remaining plasma samples (if any) will be destroyed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Biological APS: 50 Asymptomatic patients with aPL antibodies and prolonged APTT
  Interventions: Biological: blood sample
- Obstetrical APS: 50 patients with Obstetrical aPL syndrome
  Interventions: Biological: blood sample
- Thrombosis APS: APS with a personal history of venous or arterial thrombosis (50 patients)
  Interventions: Biological: blood sample

INTERVENTIONS:
Biological: blood sample — A single 15 mL blood draw is planned for this study, as follow:
  * 10 mL citrated tube (2 tubes) for APTT, PT, D-Dimers, LA, aCL, aβ2GP1, aβ2GP1-dm1 and TGA
  * 5 mL EDTA tube for blood count
  During a follow up visit, a 5 ml citrated tube and a 5 mL EDTA tube are collected from each patient for their routine laboratory evaluation. One additional citrated tube will be required to measure thrombin generation and aβ2GP1-dm1.

SUMMARY:
Antiphospholipid syndrome (APS) is an autoimmune disease characterized by thromboembolic events or pregnancy complications associated with circulating antiphospholipid antibodies (aPL-Abs). APS diagnosis needs the presence of both clinical and serological criteria (SAPORRO criteria, updated with Sydney criteria in 2006). However, no correlation between laboratory assays and the clinical thrombosis risk in patients with aPL-Abs was observed as only few patients with aPL-Abs developed clinical manifestations. Thrombin generation assays (TGA) is a global coagulation test that may represent a certain interest to evaluate thrombosis risk as a high thrombin generation capacity seems to be an independent risk factor for recurrent thromboembolic events. Another point of interest to assess the thrombotic risk is the detection of autoantibodies recognizing domain 1 of β2Gp1 (aβ2GP1-dm1). These autoantibodies are strongly related correlated with thrombotic and pregnancy manifestations. Recently, a commercial chemiluminescence immunoassay (CLIA) for detection of aβ2GP1-dm1 became available on Acustar® analyzer (HemosIL Acustar®, Instrument Laboratory, Bedford, USA) to facilitate aβ2GP1-dm1 research.

The aim of this study is to evaluate two additional laboratory assays to improve the correlation between laboratory assays and the clinical thrombosis risk in patients with antiphospholipid (APL): thrombin generation assay and aβ2GP1-dm1. Each biological result (Antibodies to Domain 1 (Dm1) of β2-Glycoprotein 1 (aβ2GP1-dm1) and Thrombin Generation Test (TGT) parameters: endogen thrombin potential (ETP), lag time and time to peak) will be compared to the history of clinical thrombosis (venous or arterial thrombosis and/or obstetrical complications such as defined by the Saporro criteria updated with Sydney criteria in 2006) for each patient.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with confirmed aPL-Abs (at least two positive determinations at least 12 week apart)
* Subject non opposition

Exclusion Criteria:

* Age < 18 years
* Patient under the protection of justice, under guardianship or under curatorship
* Patient with anticoagulant treatment, except heparin
* Clinically symptomatic liver disease, supported by e.g. diagnosis of cirrhosis, portal hypertension, ascites, PT superior or egal to 5 seconds above upper normal limit
* Platelet count < 100 G/L (giga/liter)
* Poor venous access
* Non confirmed suspicion of APS

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 150 adult patients with known aPL-Abs (Antiphospholipid antibodies) will be including in the study after collecting their informed consent.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2019-03-13 (Actual); Primary Completion 2027-03-13 (Estimated); Study Completion 2027-03-13 (Estimated)

PRIMARY OUTCOMES:
aβ2GP1-dm | One day
  The hypercoagulability status will be compared in each group. Each biological result of aβ2GP1-dm1 will be compared to a gold standard: the history of clinical thrombosis (venous or arterial thrombosis and/or obstetrical complications such as defined by the Saporro criteria updated with Sydney criteria in 2006) for each patient.
Endogenous Thrombin Potential (ETP) | One day
  The hypercoagulability status will be compared in each group. Each biological result of ETP will be compared to a gold standard: the history of clinical thrombosis (venous or arterial thrombosis and/or obstetrical complications such as defined by the Saporro criteria updated with Sydney criteria in 2006) for each patient.
peak of thrombin | One day
  The hypercoagulability status will be compared in each group. Each biological result of peak of thrombin will be compared to a gold standard: the history of clinical thrombosis (venous or arterial thrombosis and/or obstetrical complications such as defined by the Saporro criteria updated with Sydney criteria in 2006) for each patient.
lag time | One day
  The hypercoagulability status will be compared in each group. Each biological result of lag time will be compared to a gold standard: the history of clinical thrombosis (venous or arterial thrombosis and/or obstetrical complications such as defined by the Saporro criteria updated with Sydney criteria in 2006) for each patient.
time to peak | One day
  The hypercoagulability status will be compared in each group. Each biological result of time to peak will be compared to a gold standard: the history of clinical thrombosis (venous or arterial thrombosis and/or obstetrical complications such as defined by the Saporro criteria updated with Sydney criteria in 2006) for each patient.

CONTACTS AND LOCATIONS:
Locations (4):
- France (4):
  - Hôpital Cardiologique Louis Pradel, Bron
  - CHU de Clermont-Ferrand, Clermont-Ferrand
  - Hôpital Edouard Herriot, Lyon
  - Centre Hospitalier Lyon Sud, Pierre-Bénite